CLINICAL TRIAL: NCT00539474
Title: "The Efficacy of 'Radioguided Occult Lesion Localization' (ROLL) Versus 'Wire-guided Localization' (WGL) in Breast Conserving Surgery for Non-palpable Breast Cancer: a Randomized Clinical Trial"
Acronym: ROLL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, R. van Hillegersberg, Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/089; ZonMw grant: 80-82310-98-08004
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: ROLL trial; Minimally invasive surgery; Non palpable breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Wireguided localisation
  Interventions: Procedure: Radio guided occult lesion localisation
- 2 (Experimental): Radioguided occult lesion localisation
  Interventions: Procedure: Radio guided occult lesion localisation

INTERVENTIONS:
Procedure: Radio guided occult lesion localisation — ROLL procedure using the Europrobe (Europrobe, Strassbourg, France) WGL using a hook wire

SUMMARY:
Rationale:

Approximately 25% of breast cancers detected are non palpable. Accordingly, a localization technique is required to help the surgeon to find and remove the cancer. The current technique (wire guided localization [WGL]) is difficult to perform and has a high rate of tumour positive margins in the resected specimen, requiring a second operation. A new approach in the localization and resection of non-palpable malignant breast lesions is 'radio guided occult lesion localization' (ROLL). ROLL was introduced as a possible replacement for WGL at the 'European Institute of Oncology' in Milan in 1996. This technique utilizes the intratumourally injected radiotracer, that is generally used for the lymphatic mapping and SNB, to localize the primary tumour guided by the gamma probe. Five studies so far have proven the applicability of this method.

Objective:

To evaluate the efficacy of Radio Occult Lesion Localisation (ROLL) versus Wire guided Localisation (WGL) in breast conserving surgery for non-palpable breast cancer

Study design:

A multicenter, prospective randomized clinical trial. Patients with proven non-palpable breast cancer will be randomized for either ROLL or WGL.

Study population:

316 women with a core biopsy proven non palpable cT1 breast carcinoma that are eligible for a breast conserving treatment and sentinel node biopsy (SNB).

Intervention (if applicable):

Patients in the WGL group will undergo intra tumoural injection of a nuclear radiotracer under stereotactic or ultrasonographic guidance. After scintigraphic imaging, to monitor the migration of the radiotracer, a guide wire will be inserted under stereotactic or ultrasonographic guidance. The excision of the primary tumour is guided by the inserted wire and the sentinel node procedure is performed using a gamma probe and intratumoural injection of patent blue.

Patients in the ROLL group will undergo the same procedure except for the guide wire insertion. The excision of the primary tumour is guided by the gamma probe.

Main study parameters/endpoints:

Primary study endpoints; ROLL vs WGL:

1. The percentage of tumour-free margins (invasive and in situ)
2. The volume and maximum diameter of the lumpectomy

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

There is no pre-, per- or post operative extra burden. The radiofarmacon is already used in the standard care of breast cancer patients for the sentinel node biopsy. The used radio-active substance does not damage the patient.

A specific burden questionnaire, aimed at evaluating the burden of the cosmetic result, will be administered. To further assess the net impact in terms of Health Related Quality of Life (HRQoL) also the EQ5D will be obtained at T = 0, 6, 12 and 26 weeks after the initial diagnostic work-up.

Should the results indicate that overall the WGL procedure lead to better clinical outcome a cost-effectiveness analysis is foreseen using bootstrapping to assess the uncertainty with regard to the balance between costs and effects. All analyses will be limited to a half year time horizon. Accordingly, discounting of costs or effects is not applicable.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years, with a non-palpable breast carcinoma (cT1) that need to be treated with a lumpectomy and sentinel node biopsy

Exclusion Criteria:

* Pregnant patients or patients who breast feed
* Patients with multi focal tumour growth
* Patients with only ductal carcinoma in situ or lobular carcinoma in situ in the core biopsy
* Patients requiring breast amputation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Radicality, oncologic outcome | 3 years

SECONDARY OUTCOMES:
Doctors questionnaires Patients questionnaire cost-effectiveness analysis | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: R van Hillegersberg, dr, Principal Investigator — UMCU
Locations (4):
- Netherlands (4):
  - Amphia hospital, Breda, North Brabant
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - st Antonius Hospital, Nieuwegein, Utrecht
  - University Medical Center, Utrecht, Utrecht

REFERENCES:
- [Derived] Postma EL, Koffijberg H, Verkooijen HM, Witkamp AJ, van den Bosch MA, van Hillegersberg R. Cost-effectiveness of radioguided occult lesion localization (ROLL) versus wire-guided localization (WGL) in breast conserving surgery for nonpalpable breast cancer: results from a randomized controlled multicenter trial. Ann Surg Oncol. 2013 Jul;20(7):2219-26. doi: 10.1245/s10434-013-2888-7. Epub 2013 Feb 23. PMID 23435568
- [Derived] Postma EL, Verkooijen HM, van Esser S, Hobbelink MG, van der Schelling GP, Koelemij R, Witkamp AJ, Contant C, van Diest PJ, Willems SM, Borel Rinkes IH, van den Bosch MA, Mali WP, van Hillegersberg R; ROLL study group. Efficacy of 'radioguided occult lesion localisation' (ROLL) versus 'wire-guided localisation' (WGL) in breast conserving surgery for non-palpable breast cancer: a randomised controlled multicentre trial. Breast Cancer Res Treat. 2012 Nov;136(2):469-78. doi: 10.1007/s10549-012-2225-z. Epub 2012 Sep 30. PMID 23053639
- [Derived] van Esser S, Hobbelink MG, Peeters PH, Buskens E, van der Ploeg IM, Mali WP, Rinkes IH, van Hillegersberg R. The efficacy of 'radio guided occult lesion localization' (ROLL) versus 'wire-guided localization' (WGL) in breast conserving surgery for non-palpable breast cancer: a randomized clinical trial - ROLL study. BMC Surg. 2008 May 21;8:9. doi: 10.1186/1471-2482-8-9. PMID 18495027